CLINICAL TRIAL: NCT06797791
Title: Multifocal Theta Burst Transcranial Magnetic Stimulation in Generalized Epilepsy Management.
Brief Title: Assessment of Multifocal Continuous Theta Burst Transcranial Magnetic Stimulation (cTBS) Effects in Generalized Epilepsy Patients.
Acronym: TBS-GEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitatea de Stat de Medicina si Farmacie Nicolae Testemiţanu (Other)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Pavel Leahu, Dr., Asst. prof., PhD candidate, Universitatea de Stat de Medicina si Farmacie Nicolae Testemiţanu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19062018-85
Record Dates: First submitted 2024-11-03; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Generalized Epilepsy
Keywords: TBS; cTBS; IGE; Generalized; Epilepsy; Theta; Burst; Transcranial; Magnetic; Stimulation; Continuous
MeSH Terms: conditions — Epilepsy, Generalized; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multifocal continuous theta burst transcranial magnetic stimulation (Experimental): After determining the resting motor threshold (RMT), all subjects underwent 6 sessions of continuous theta burst stimulation (cTBS) for 6 consecutive days according to the research protocol. TBS sessions were accompanied by parallel high-density electroencephalography (hdEEG) monitoring. Afterward, a follow-up period of up to three months with visits at predefined intervals of 4, 8, and 12 weeks was carried out.
  Interventions: Device: Multifocal Continuous Theta Burst Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Multifocal Continuous Theta Burst Transcranial Magnetic Stimulation — The experimental stimulation protocol included 3 trains of cTBS with an inter-train interval of 10 min. Each train of cTBS consisted of 600 pulses applied in blocks at the theta frequency (200ms) with a duration of 40 s. A block of pulses consisted of 3 pulses at 50Hz frequency, stimulus intensity being estimated as 80% of the RMT. Stimulation application was performed by positioning the Magventure MMC-140 coil over the vertex (Cz) according to the 10-20 EEG system overlapping bilateral motor and somatosensory cortical areas.
  Other Names: cTBS

SUMMARY:
The goal of this clinical study is to assess the efficacy of multifocal theta burst transcranial magnetic stimulation in the prevention of epileptic seizures in adult patients with generalized epilepsy. The main questions it aims to answer are:

* How does multifocal continuous theta burst stimulation (cTBS) impact the frequency and severity of epileptic seizures?
* Does cTBS influence the quality of life in patients with generalized epilepsy?
* What is the safety and tolerability profile of the experimental multifocal cTBS protocol?

ELIGIBILITY:
Inclusion Criteria:

- Adult patients with generalized epilepsy (according to ILAE 2017 classification of epilepsy).

Exclusion Criteria:

* refusal to sign the informed consent;
* focal, combined or unknown epilepsy (according to ILAE criteria);
* drug-resistant form of epilepsy (according to ILAE definition);
* history or symptoms of renal or hepatic failure;
* history of oncological disorder;
* uncontrolled high blood pressure;
* cognitive impairment;
* psychiatric disorders;
* signs of structural brain injury or focal neurological symptoms;
* use of opioids or muscle relaxants;
* history of substance abuse;
* ferromagnetic implants in head and neck regions;
* cardiac pacemakers;
* pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Seizure frequency | at 12 weeks
  ≥50% improvement from Baseline in seizure frequency

SECONDARY OUTCOMES:
Quality of Life in Epilepsy (QOLIE-31) Inventory | at 12 weeks
  Exploratory analyses will investigate the changes in the 31-item Quality of Life in Epilepsy (QOLIE-31) score from Baseline due to study protocol and interventions. The questionnaire comprises seven categories: worry about epileptic seizures, emotional well-being, energy/fatigue, social function, cognitive function, medication effects, and general quality of life. The scale is scored from 0 to 100. Higher scores reflect a higher quality of life.
Seizure Severity Questionnaire (SSQ) | at 12 weeks
  Exploratory analyses will investigate the changes in the Seizure Severity Questionnaire (SSQ) score from Baseline due to study protocol and intervention. The SSQ is a 24-item questionnaire that includes questions regarding the frequency and usefulness of warning signs, severity and disturbance of ictal movements, loss of consciousness, and frequency, severity, and postictal cognitive, emotional, and physical disturbance. Scores per category range from 1 to 7, with higher scores indicating greater severity.
Patient Global Impression of Change (PGIC) | at 12 weeks
  Improvement in Patient Global Impression of Change (PGIC) score from Baseline. PGIC is used to assess patients' perceptions of changes after treatment. It is a 7-point scale with the options "very much improved", "much improved", "minimally improved", "no change", "minimally worsened", "much worsened" and "very much worsened".

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From start of intervention (Day 1) through 6 consecutive days (Day 6) of treatment
  After each continuous Theta Burst Stimulation (cTBS) session an assessment of possible adverse events ( CTCAE v4.0 terms) occurring during and/or immediately after stimulation was done.

CONTACTS AND LOCATIONS:
Locations (2):
- Moldova (2):
  - Emergency Medicine Institute, Chisinau
  - Nicolae Testemițanu State University of Medicine and Pharmacy, Chisinau

IPD SHARING:
Plan to Share IPD: Undecided